CLINICAL TRIAL: NCT03015311
Title: Strategy of Systolic Blood Pressure Intervention in the Elderly Hypertensive Patients: A Prospective Randomized Open-Label Blinded-Endpoint Trial
Brief Title: Strategy of Blood Pressure Intervention in the Elderly Hypertensive Patients
Acronym: STEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Cai, Director, Hypertension Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016CXGC07; 2016-I2M-1-006 (Other Grant/Funding Number: CAMS Innovation Fund for Medical Sciences)
Record Dates: First submitted 2017-01-02; First posted 2017-01-10 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Primary Hypertension
Keywords: Blood pressure control
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive BP control (Experimental): SBP within 110 - <130 mm Hg. Participants randomized into the Intensive BP control arm will have a goal of SBP 110 - <130 mm Hg.
  Interventions: Drug: Intensive BP control
- Standard BP control (Active Comparator): SBP within 130 - <150 mm Hg. Participants randomized into the Intensive BP control arm will have a goal of SBP 130 - <150 mm Hg.
  Interventions: Drug: Standard BP control

INTERVENTIONS:
Drug: Intensive BP control — For all participants, Olmesartan Medoxomil tablets or Amlodipine Besylate tablets will be used as an initial therapy. Other drugs, including hydrochlorothiazide and β-blockers, are allowed, in order to achieve the SBP target. If the target BP level is not achieved during the Follow-up periods, adjustment of drug type and dosage will be carried out according to procedures defined in the protocol.
  Other Names: Lower target for reducing SBP
  Arms: Intensive BP control
Drug: Standard BP control — For all participants, Olmesartan Medoxomil tablets or Amlodipine Besylate tablets will be used as an initial therapy. Other drugs, including hydrochlorothiazide and β-blockers, are allowed, in order to achieve the SBP target. If the target BP level is not achieved during the Follow-up periods, adjustment of drug type and dosage will be carried out according to procedures defined in the protocol.
  Other Names: Standard target for reducing SBP
  Arms: Standard BP control

SUMMARY:
The Strategy of Blood Pressure Intervention in the Elderly Hypertensive Patients (STEP) is a 2-arm, multi-center, prospective, randomized, open-labeled, blinded-endpoint trial. The purpose of this trial is to test whether a treatment program aimed at reducing systolic blood pressure (SBP) to a lower goal (<130 mmHg, intensive treatment) than currently recommended (<150 mmHg, standard treatment) will reduce CVD risk among persons between 60-80 years of old. Furthermore, this trial will also examine the effect of blood pressure APP management strategy via WeChat network on medication compliance, blood pressure control and CVD benefits.

DETAILED DESCRIPTION:
Hypertension is highly prevalent in the adult population in China, and its burden is rapidly increasing among persons older than 60 years of age. Elevated blood pressure (BP) is an important public health concern which contributes to several adverse health outcomes, especially coronary heart disease, stroke, heart failure, chronic kidney disease, and decline in cognitive function. Clinical trials have shown that a lower systolic blood pressure goal will lead to greater reduction in cardiovascular disease (CVD) incidence, but the effect of intensive treatment of systolic blood pressure below 120 mm Hg in reducing of CVD risk has long been debated. In particularly, among the elderly hypertensive patients aged 60 years or older, the most appropriate targets for blood pressure lowering to reduce cardiovascular events still remain uncertain.

The STEP trial will randomize about 8000 participants aged between 60 and 80 years with SBP≥140 mm Hg and <190 mm Hg, and without a history of atherothrombotic or hemorrhagic stroke. Target SBP goals are 110-130 vs 130-150 mm Hg, respectively. The purpose of the STEP trial is to test whether a treatment program aimed at reducing systolic blood pressure (SBP) to a lower goal (<130 mmHg, intensive treatment) than currently recommended (<150 mmHg, standard treatment) will reduce CVD risk among hypertensive patients between 60-80 years. Participants will be recruited at approximately 40 clinic centers in China within approximately a 1-year period, and will be followed for 4 years. Furthermore, this trial will also examine the effect of blood pressure APP management strategy via WeChat network on medication compliance, blood pressure control and CVD benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Systolic BP between 140-190 mm Hg in the three screening visits or currently under anti-hypertension treatment；
2. An age of 60 - 80 years old；
3. Signed the written informed consent.

Exclusion Criteria:

1. Systolic BP≥190 mm Hg, or diastolic BP <60 mm Hg;
2. Known secondary cause of hypertension;
3. History of large atherosclerotic cerebral infarction or hemorrhagic stroke (not lacunar infarction and transient ischemic attack [TIA]);
4. Hospitalization for myocardial infarction or unstable angina within the previous 6 months;
5. Coronary revascularization (PCI or CABG) within the previous 12 months;
6. Planned to perform coronary revascularization (PCI or CABG) in the future 12 months;
7. History of sustained atrial fibrillation or Ventricular arrhythmias at entry influencing the measurement of electronic blood pressure；
8. NYHA class III-IV heart failure at entry or hospitalization for exacerbation of chronic heart failure within the previous 6 months;
9. Severe valvular disease or valvular disease likely to require surgery or percutaneous valve replacement during the trial;
10. Dilated or hypertrophic cardiomyopathy, rheumatic heart disease, or congenital heart disease;
11. Uncontrolled diabetes (serum fasting glucose ≥200 mg/dl [11.1 mmol/L], HbA1>8%);
12. Lab tests indicating abnormal liver or kidney function (ALT more than 3 times the upper limit of normal value, or end stage renal disease (ESRD) on dialysis, or estimated glomerular filtration rate (eGFR) <30 mL/min, or serum creatine >2.5 mg/dl [>221 umol/L];
13. Severe somatic disease such as cancer;
14. Severe cognitive impairment or mental disorders;
15. Participating in other clinical trials.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2017-01-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary composite outcome | 4 years
  A composite end-point comprised of acute coronary syndrome (myocardial infarction and hospitalization for unstable angina), first occurrence of symptomatic stroke ( ischemic or hemorrhagic stroke), hospitalization for decompensated heart failure, coronary revascularization (percutaneous coronary intervention [PCI], coronary artery bypass grafting [CABG]), atrial fibrillation, and death from cardiovascular causes.

SECONDARY OUTCOMES:
Composite of major adverse cardiac events (primary outcome without stroke) | 4 years
  Composite of major adverse cardiac events comprised of acute coronary syndrome (myocardial infarction and hospitalization for unstable angina), hospitalization for decompensated heart failure, coronary revascularization (percutaneous coronary intervention [PCI], coronary artery bypass grafting [CABG]), atrial fibrillation, and death from cardiovascular causes.
First occurrence of symptomatic stroke ( ischemic or hemorrhagic) | 4 years
  Stroke is defined as a rapid onset of focal (or global) disturbance of cerebral function lasting more than 24 hours (except interrupted by surgery or death) without resolution of symptoms according to the World Health Organization. The diagnosis of stroke is confirmed by strict neurological examination, computed tomography (CT), or magnetic resonance imaging (MRI), and stroke subtypes are classified including ischemic or hemorrhagic, fatal or not fatal.
Acute coronary syndrome | 4 years
  Acute coronary syndrome includes myocardial infarction and hospitalization for unstable angina. The diagnosis of MI is based on the following criteria: (1) Patient has cardiac signs and symptoms, such as retrosternal pain last for at least 30 minutes, and not relieve to nitroglycerine during the attack; (2) Electrocardiographic abnormal findings of MI are observed; (3) Biochemical markers of cardiac damage are present.
  The diagnosis of unstable angina requires hospitalization for evaluation. The clinical presentation of unstable angina includes: (1) prolonged (>20 min) angina pain at rest; (2) new onset angina; (3) post-MI angina; (4) recent destabilization of previously stable angina with at least Canadian Cardiovascular Society Class III angina characteristics.
Hospitalization for acute decompensated heart failure | 4 years
  Diagnosis of acute decompensated heart failure requires a hospitalization or emergency department visit which provides an infusion therapy for clinical signs and symptoms consistent with cardiac decompensation or inadequate cardiac pump function, such as increasing or new onset shortness of breath, peripheral edema, paroxysmal dyspnea, orthopnea, or hypoxia.
coronary revascularization (percutaneous coronary intervention [PCI], coronary artery bypass grafting [CABG]) | 4 years
  Patients are treated with coronary revascularization by either PCI or CABG due to acute coronary syndromes (ACS) and stable ischemic heart disease (SIHD).
Atrial fibrillation | 4 years
  Diagnosis of AF requires rhythm evidence of an ECG showing the typical pattern including absolutely irregular RR intervals and no discernible, distinct P waves.
Cardiovascular death | 4 years
  Cardiovascular death includes fatal coronary heart disease, fatal stroke, death from heart failure, and sudden cardiac death.
All-cause death | 4 years
  All-cause death includes death due to any reasons during the trial. Evidence for death includes death certificates from hospitals or reports of home visit from investigators.
First occurrence of diabetes mellitus | 4 years
  Diagnosis of incident diabetes mellitus includes the following criteria: (1) Fasting plasma glucose ≥ 126 mg/dl (≥ 7.0 mmol/dl); or (2) Oral glucose tolerance test 2-hour glucose in venous plasma ≥ 200 mg/dl (≥ 11.1 mmol/l); or (3) In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥ 200 mg/dl (≥ 11.1 mmol/l); or (4) Glycosylated hemoglobin (HbA1c) ≥ 6.5% (48 mmol/mol).
Decline in cognitive function | 4 years
  Decline in cognitive function includes sensory disturbance, memory disorders and thinking disorders, which is assessed by mini-mental state examination (MMSE)
Decline in renal function or development of end stage renal disease (ESRD) | 4 years
  Decline in renal function is assessed by any of the following: (1) For patients with chronic kidney disease (eGFR <60 ml per minute per 1.73 m2) at baseline, the renal outcome was a composite of a decrease in the eGFR of 50% or more (confirmed by a subsequent laboratory test) or the development of ESRD requiring long-term dialysis or kidney transplantation; or (2) For participants without chronic kidney disease at baseline, the renal outcome was defined by a decrease in the eGFR of 30% or more to a value of less than 60 ml per minute per 1.73 m2.
Major artery stiffness | 4 years
  Major artery stiffness are assessed by a composite of decrease in the ankle brachial index [ABI], brachial-ankle pulse wave velocity(baPWV), or brachial artery flow-mediated dilation [FMD].
  ABI and baPWV,well-established non-invasive techniques for evaluating obstruction and stiffness of peripheral artery respectively, are considered for the purposes of cardiovascular risk assessment. ABI is the ratio of the average systolic blood pressure measured in brachial/ankle, and an ABI between and including 0.9 and 1.2 is considered normal, while a lesser than 0.9 indicates arterial disease. The unit measure of baPWV value is cm per second.
  FMD serves as an index of nitric oxide (NO)-mediated endothelium-dependent vasodilator function in humans and is regarded as a surrogate marker of cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, MD, Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (42):
- China (42):
  - Beijing Chaoyang Hospital affiliated to Capical Medical University, Beijing, Beijing Municipality
  - Bei Jing Hospital, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences, FuWai Hospital, Beijing, Beijing Municipality
  - Xuanwu hospital of capital medical university, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong Cardiovascular Institute, Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - The Second Affiliated Hospital to Medical College Shantou University Guangdong, Shantou, Guangdong
  - Shenzhen Sun Yat-sen Cardiovascular Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi
  - Kailua General Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - First affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hong xinglong center hospital, Shuangyashan, Heilongjiang
  - First Affiliated Hospitalof Zhengzhou University, Zhengzhou, Henan
  - Zhoukou City Central Hospital, Zhoukou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Kang Ya Hospita, Yiyang, Hunan
  - The Second Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Zhenjiang First People's Hospital, Zhenjiang, Jiangsu
  - the Second Affiliated Hospitalof NanChang University, Nanchang, Jiangxi
  - Benxi Railway Hospital, Benxi, Liaoning
  - The 1st Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Shanghai general hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi caidiovascular hospital, Taiyuan, Shanxi
  - Shanxi Academy of Medical Sciences, Shanxi Dayi Hospital, Taiyuan, Shanxi
  - First Affiliated Hospital, Xian Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - College of Medicine , National Taiwan University, Taibei, Taiwan
  - Pingjin Hospital, Logistics University of PAPF, Tianjin, Tianjin Municipality
  - the People's Hospital of Ji Xian Distric, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yan'an Hospital affiliated to kunming medical university, Yunnan Cardiovascular Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Hospital of Kunming, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
Within 3 years after the trial complete
Supporting Information: Study Protocol, SAP
Time Frame: Within 3 years after the trial complete
Access Criteria: To share IPD in the magazine of paper published

REFERENCES:
- [Background] Wang Y, Peng X, Nie X, Chen L, Weldon R, Zhang W, Xiao D, Cai J. Burden of hypertension in China over the past decades: Systematic analysis of prevalence, treatment and control of hypertension. Eur J Prev Cardiol. 2016 May;23(8):792-800. doi: 10.1177/2047487315617105. Epub 2015 Nov 24. PMID 26603746
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] ACCORD Study Group; Cushman WC, Evans GW, Byington RP, Goff DC Jr, Grimm RH Jr, Cutler JA, Simons-Morton DG, Basile JN, Corson MA, Probstfield JL, Katz L, Peterson KA, Friedewald WT, Buse JB, Bigger JT, Gerstein HC, Ismail-Beigi F. Effects of intensive blood-pressure control in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1575-85. doi: 10.1056/NEJMoa1001286. Epub 2010 Mar 14. PMID 20228401
- [Background] Probstfield JL, Applegate WB, Borhani NO, Curb JD, Cutler JA, Davis BR, Furberg CD, Hawkins CM, Lakatos E, Page LB, et al. The Systolic Hypertension in the Elderly Program (SHEP): an intervention trial on isolated systolic hypertension. SHEP Cooperative Research Group. Clin Exp Hypertens A. 1989;11(5-6):973-89. doi: 10.3109/10641968909035386. PMID 2676266
- [Background] JATOS Study Group. Principal results of the Japanese trial to assess optimal systolic blood pressure in elderly hypertensive patients (JATOS). Hypertens Res. 2008 Dec;31(12):2115-27. doi: 10.1291/hypres.31.2115. PMID 19139601
- [Derived] Song Q, Peng X, Bai J, Yang R, Ling Q, Chen S, Ji Y, Dong X, Wang X, Wu S, Wang TD, Yu X, Liu H, Ren J, Zhou X, Chen R, Yang L, Yang J, Tian G, Zhang H, Zhao D, Chen F, Li D, Yu J, Zhang J, Yang Z, Zhang W, Cai J. Intensive Blood Pressure Control in Older Patients With Hypertension: 6-Year Results of the STEP Trial. J Am Coll Cardiol. 2025 Oct 28;86(17):1421-1433. doi: 10.1016/j.jacc.2025.06.045. Epub 2025 Oct 17. PMID 41105077
- [Derived] Ji Y, Peng X, Chen S, Song Q, Bai J, Cai J. Evening home pulse pressure predicted cardiovascular events and mortality in older adults with hypertension: findings based on the STEP trial. Hypertens Res. 2025 Nov;48(11):2801-2810. doi: 10.1038/s41440-025-02349-y. Epub 2025 Aug 26. PMID 40858751
- [Derived] Dong X, Bai J, Ling Q, Zhao X, Cai J. Effect of Intensive Blood Pressure Control in Patients with Resistant Hypertension: Insights from the STEP Trial. Eur J Prev Cardiol. 2025 Aug 12:zwaf507. doi: 10.1093/eurjpc/zwaf507. Online ahead of print. PMID 40796327
- [Derived] Peng X, Olsen MH, Pareek M, Bai J, Liu Y, Song Q, Cai J. Impact of antihypertensive drug classes on cardiovascular outcomes: insights from the STEP study. BMC Med. 2025 Jul 1;23(1):365. doi: 10.1186/s12916-025-04158-z. PMID 40598287
- [Derived] Ling Q, Dong X, Bai J, Deng Y, Song Q, Cai J. Impact of Hypertension Duration on the Cardiovascular Benefit of Intensive Blood Pressure Control. Hypertension. 2024 Sep;81(9):1945-1955. doi: 10.1161/HYPERTENSIONAHA.124.23439. Epub 2024 Jul 17. PMID 39016010
- [Derived] Zhang K, Song Q, Bai J, Cai J. Association of intensive blood pressure management with cardiovascular outcomes in patients using multiple classes of antihypertensive medications: a post-hoc analysis of the STEP Trial. Hypertens Res. 2024 Jul;47(7):1779-1788. doi: 10.1038/s41440-024-01647-1. Epub 2024 Apr 10. PMID 38600278
- [Derived] Zhao S, Deng Y, Wang Y, Yu S, Han J, Cai J, Zhang Y. Incidence and prognosis of cardiac conduction system diseases in hypertension: the STEP trial. Nat Aging. 2024 Apr;4(4):483-490. doi: 10.1038/s43587-024-00591-6. Epub 2024 Mar 21. PMID 38514823
- [Derived] Yang R, Zhang J, Yu X, Yang G, Cai J. Remnant cholesterol and intensive blood pressure control in older patients with hypertension: a post hoc analysis of the STEP randomized trialdagger. Eur J Prev Cardiol. 2024 Jun 3;31(8):997-1004. doi: 10.1093/eurjpc/zwae001. PMID 38167928
- [Derived] Zhang S, Zhong Y, Wu S, Wu H, Cai J, Zhang W; STEP Study Group. Intensive blood pressure control on arterial stiffness among older patients with hypertension. Chin Med J (Engl). 2024 May 5;137(9):1078-1087. doi: 10.1097/CM9.0000000000002868. Epub 2023 Nov 15. PMID 37968125
- [Derived] Yang R, Huang R, Zhang L, Li D, Luo J, Cai J. Influence of Baseline Diastolic Blood Pressure on the Effects of Intensive Blood Pressure Lowering: Results From the STEP Randomized Trial. Hypertension. 2023 Dec;80(12):2572-2580. doi: 10.1161/HYPERTENSIONAHA.123.21892. Epub 2023 Oct 10. PMID 37814892
- [Derived] Gonzalez-Vilchez F, Hernandez-Perez F, Almenar-Bonet L, Crespo-Leiro MG, Lopez-Granados A, Ortiz-Bautista C, Delgado-Jimenez JF, de Antonio-Ferrer M, Sobrino-Marquez JM, Garcia-Romero E; Spanish Heart Transplant Teams. Spanish heart transplant registry. 34th official report of the Heart Failure Association of the Spanish Society of Cardiology. Rev Esp Cardiol (Engl Ed). 2023 Nov;76(11):901-909. doi: 10.1016/j.rec.2023.06.013. Epub 2023 Sep 6. English, Spanish. PMID 37683823
- [Derived] Wang X, Feng Y, Yang L, Zhang G, Tian X, Ling Q, Tan J, Cai J. Association of baseline serum cholesterol with benefits of intensive blood pressure control. Chin Med J (Engl). 2023 Sep 5;136(17):2058-2065. doi: 10.1097/CM9.0000000000002474. PMID 37525354
- [Derived] Deng Y, Bai J, Yang X, Liu W, Guo Z, Zhang J, Huang R, Yang X, Yu C, Yu J, Guo X, Wu H, Liu P, Zhang W, Cai J. Achieved systolic blood pressure and cardiovascular outcomes in 60-80-year-old patients: the Strategy of Blood Pressure Intervention in the Elderly Hypertensive Patients (STEP) trial. Eur J Prev Cardiol. 2023 Aug 1;30(10):1017-1027. doi: 10.1093/eurjpc/zwad142. PMID 37172116
- [Derived] Yu J, Song Q, Bai J, Wu S, Bu P, Li Y, Cai J. Visit-to-Visit Blood Pressure Variability and Cardiovascular Outcomes in Patients Receiving Intensive Versus Standard Blood Pressure Control: Insights From the STEP Trial. Hypertension. 2023 Jul;80(7):1507-1516. doi: 10.1161/HYPERTENSIONAHA.122.20376. Epub 2023 May 12. PMID 37170806
- [Derived] Yang R, Zhu Y, Xu M, Tao Y, Cong W, Cai J. Intensive blood pressure lowering and the risk of new-onset diabetes in patients with hypertension: a post-hoc analysis of the STEP randomized trial. Eur J Prev Cardiol. 2023 Aug 1;30(10):988-995. doi: 10.1093/eurjpc/zwad105. PMID 37036035
- [Derived] Fan J, Bai J, Liu W, Cai J. Effects of intensive vs. standard blood pressure control on cognitive function: Post-hoc analysis of the STEP randomized controlled trial. Front Neurol. 2023 Feb 1;14:1042637. doi: 10.3389/fneur.2023.1042637. eCollection 2023. PMID 36816574
- [Derived] Wang XQ, Tan JS, Zhang SY, Zhang WL, Cai J. Association of serum uric acid with benefits of intensive blood pressure control. Rev Esp Cardiol (Engl Ed). 2023 Aug;76(8):635-644. doi: 10.1016/j.rec.2023.01.003. Epub 2023 Jan 28. English, Spanish. PMID 36716991
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Ling Q, Song Q, Bai J, Wu S, Zhang W, Chen M, Cai J. Temporal Relationship Between Arterial Stiffness and Systolic Blood Pressure Under Intensive or Standard Control: A Post Hoc Analysis of the STEP Trial. Hypertension. 2022 Dec;79(12):2755-2763. doi: 10.1161/HYPERTENSIONAHA.122.20022. Epub 2022 Oct 24. PMID 36278416
- [Derived] Song Q, Ling Q, Bai J, Zhang H, Bu P, Chen F, Wu S, Zhang W, Chen M, Cai J. Influence of baseline arterial stiffness on effects of intensive compared with standard blood pressure control: a post hoc analysis of the STEP trial. BMC Med. 2022 Oct 20;20(1):358. doi: 10.1186/s12916-022-02556-1. PMID 36261812
- [Derived] Fan J, Zheng W, Liu W, Xu J, Zhou L, Liu S, Bai J, Qi Y, Huang W, Liu K, Cai J. Cost-Effectiveness of Intensive Versus Standard Blood Pressure Treatment in Older Patients With Hypertension in China. Hypertension. 2022 Nov;79(11):2631-2641. doi: 10.1161/HYPERTENSIONAHA.122.20051. Epub 2022 Sep 30. PMID 36177835
- [Derived] Zhang S, Zhong Y, Wang L, Yin X, Li Y, Liu Y, Dai Q, Tong A, Li D, Zhang L, Li P, Zhang G, Huang R, Liu J, Zhao L, Yu J, Zhang X, Yang L, Cai J, Zhang W; STEP Study Group. Anxiety, home blood pressure monitoring, and cardiovascular events among older hypertension patients during the COVID-19 pandemic. Hypertens Res. 2022 May;45(5):856-865. doi: 10.1038/s41440-022-00852-0. Epub 2022 Jan 21. PMID 35064249
- [Derived] Zhang W, Zhang S, Deng Y, Wu S, Ren J, Sun G, Yang J, Jiang Y, Xu X, Wang TD, Chen Y, Li Y, Yao L, Li D, Wang L, Shen X, Yin X, Liu W, Zhou X, Zhu B, Guo Z, Liu H, Chen X, Feng Y, Tian G, Gao X, Kario K, Cai J; STEP Study Group. Trial of Intensive Blood-Pressure Control in Older Patients with Hypertension. N Engl J Med. 2021 Sep 30;385(14):1268-1279. doi: 10.1056/NEJMoa2111437. Epub 2021 Aug 30. PMID 34491661
- [Derived] Zhang S, Zhou X, Chen Y, Wang L, Zhu B, Jiang Y, Bu P, Liu W, Li D, Li Y, Tao Y, Ren J, Fu L, Li Y, Shen X, Liu H, Sun G, Xu X, Bai J, Zhang W, Cai J; STEP Study Group. Changes in Home Blood Pressure Monitored Among Elderly Patients With Hypertension During the COVID-19 Outbreak: A Longitudinal Study in China Leveraging a Smartphone-Based Application. Circ Cardiovasc Qual Outcomes. 2021 May;14(5):e007098. doi: 10.1161/CIRCOUTCOMES.120.007098. Epub 2021 May 18. PMID 34003685
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623
- [Derived] Zhang S, Wu S, Ren J, Chen X, Zhang X, Feng Y, Zhou X, Zhu B, Yang J, Tian G, Jiang Y, Guo Z, Li Y, Wang TD, Kario K, Zhang W, Cai J; STEP Study Group. Strategy of blood pressure intervention in the elderly hypertensive patients (STEP): Rational, design, and baseline characteristics for the main trial. Contemp Clin Trials. 2020 Feb;89:105913. doi: 10.1016/j.cct.2019.105913. Epub 2019 Dec 12. PMID 31838255